CLINICAL TRIAL: NCT04918186
Title: An Immunotherapy Platform Study in Platinum Resistant High Grade Serous Ovarian Cancer
Brief Title: Immunotherapy Platform Study in Platinum Resistant High Grade Serous Ovarian Cancer
Acronym: IPROC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Cancer Research Institute, New York City (Other); AstraZeneca (Industry); BioAtla, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I240
Record Dates: First submitted 2021-05-26; First posted 2021-06-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — durvalumab; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Durvalumab + BA3011 (Arm Closed) (Experimental)
  Interventions: Drug: Durvalumab; Drug: BA3011
- Durvalumab + BA3021 (Arm Closed) (Experimental)
  Interventions: Drug: Durvalumab; Drug: BA3021
- ENB-003 + Toripalimab (Experimental)
  Interventions: Drug: ENB003; Drug: Toripalimab

INTERVENTIONS:
Drug: Durvalumab — 1500mg IV, 60 min day 1 every 4 weeks
  Arms: Durvalumab + BA3011 (Arm Closed); Durvalumab + BA3021 (Arm Closed)
Drug: BA3011 — IV
  Arms: Durvalumab + BA3011 (Arm Closed)
Drug: BA3021 — IV
  Arms: Durvalumab + BA3021 (Arm Closed)
Drug: ENB003 — IV
  Arms: ENB-003 + Toripalimab
Drug: Toripalimab — IV
  Arms: ENB-003 + Toripalimab

SUMMARY:
This study is being done to answer the following question: What are the effects of a new drug or drugs on ovarian cancer? The pre-study screening may be done to test a sample of tissue for biomarkers to determine participation in the study.

DETAILED DESCRIPTION:
This study is being conducted to determine if this approach is better or worse than the standard of care for ovarian cancer. The standard of care is defined as care most people get for ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll women with platinum resistant high grade serous ovarian cancer.
* This study is open to minorities as appropriate but is not designed to measure differences in intervention effects.
* All patients must be registered for screening prior to study enrollment, however, if biomarker testing results are not required prior to enrollment to a substudy, then enrollment can proceed immediately. CCTG will advise sites when biomarker testing results are required prior to substudy enrollment.

Additional Criteria To Be Met Prior To Sub-study Enrollment All patients must fulfill all of the following criteria to be eligible for enrollment to the study. Additional eligibility criteria and relevant timings that are specific to a substudy are listed in each substudy specific protocol.

* Patients must have platinum resistant high grade serous carcinoma of ovarian, fallopian tube or peritoneal origin defined as progression within 6 months of last platinum containing chemotherapy. Histological confirmation of the original primary tumour is required.
* All patients must have measurable disease as defined by RECIST 1.1. The criteria for defining measurable disease are as follows:

  * Chest x-ray ≥ 20 mm
  * CT scan (with slice thickness of 5 mm) ≥ 10 mm - longest diameter
  * Physical exam (using calipers) ≥ 10 mm
  * Lymph nodes by CT scan ≥ 15 mm - measured in short axis
* Patients must have at least one disease site amendable to pre and on-treatment biopsies and must consent to undergo these tumour biopsies.
* Prior surgery is permitted provided that a minimum of at least 28 days have elapsed between any major surgical procedure and date of enrollment, and that wound healing has occurred.
* Systemic Therapy:

  * There is no limit to the number of prior regimens for platinum-sensitive disease. However, patients may not have received more than one cytotoxic chemotherapy regimen for platinum-resistant disease.
  * Patients may have received non-cytotoxic therapies (excluding agents targeted by the planned substudy). Refer to each substudy protocol for exclusions.
  * Prior treatment with an immune checkpoint inhibitor (ICI) is permissible providing the ICI was not discontinued for severe or recurrent severe toxicity (including myocarditis, or other myocardiotoxicity, encephalitis, colitis, diarrhea, pancreatitis, hypo/hyper thyroidism, hypopituitarism, adrenal insufficiency, rash, autonomic neuropathy, myasthenia gravis, Guillain-Barre, myositis/polymyositis, hepatitis, nephritis, Type 1 diabetes, thrombocytopenia)
  * A minimum of 4 weeks must have elapsed between last dose of prior therapy and enrollment.
  * All reversible prior toxicity must have recovered to grade ≤ 1 (consult CCTG in the case of irreversible toxicity)
* Other Therapy:

  • Radiation, endocrine therapy, or other non-anti-cancer investigational agents are permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose and enrollment. Exceptions may be made for low-dose, non-myelosuppressive radiotherapy after consultation with CCTG.
* ECOG performance status 0 or 1 and have a life expectancy ≥ 3 months.
* Patients must be ≥ 18 years of age.
* All patients must have consented to:

  1. Release of tumour block from their primary or metastatic tumour, if available. If archival tissue is unavailable, a tumour biopsy is required during screening. The centre/pathologist must have agreed to the submission of the specimen(s).
  2. Pre and on treatment tumour biopsies:
* Core needle (a minimum of 6 core samples are required) or excisional biopsies or resected tissue specimens are required.
* CCTG will advise sites when biomarker testing results are required prior to enrollment
* Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the trial.
* Patients must have adequate organ and marrow function measured within 7 days prior to enrollment including;
* Absolute neutrophils ≥ 1.5 x 10^9/L (1500/µL)
* Platelets ≥ 100 x 10^9/L (100 x 103/µL)
* Hemoglobin ≥90g/L* (10.0 g/dL) with no blood transfusions in the past 28 days.
* Bilirubin ≤ 1.5 x ULN (upper limit of normal)**
* AST & ALT ≤ 2.5 x ULN; if patient has liver metastases ≤ 5.0 x ULN
* Serum creatinine or: Creatinine clearance ≤ 1.5 x ULN / >50 mL/min
* Albumin >35 g/L (3.5 g/dL)
* INR/PTT INR < 1.7 or PTT < 4 seconds above control
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow up. Patients enrolled on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial.
* Patient must agree to return to their primary care facility for any adverse events, response assessments and follow-up, which may occur through the course of the trial.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient enrollment.
* Women of childbearing potential will have a pregnancy test to determine eligibility as part of the Pre-Study Evaluation

Exclusion Criteria:

* Patients with a history of other malignancy may be eligible if curatively treated and/or the malignancy does not affect the determination of safety or efficacy of the investigational regimen (must be confirmed with CCTG prior to enrollment).
* Patients with uncontrolled or serious illnesses, or medical conditions which could cause unacceptable safety risks or would not permit the patient to be managed according to the protocol or substudy. This includes but is not limited to:

  * history of intra-abdominal abscess within 3 months prior to starting treatment;
  * other active infection or chronic liver disease requiring systemic therapy;
  * active or known human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection on antiviral treatment or with detectable viral load;
  * history of interstitial lung disease, non-infectious pneumonitis or severe pulmonary disease exacerbated by pneumonitis or uncontrolled diseases, including pulmonary fibrosis, acute lung disease, etc.
  * clinically significant pleural, pericardial, and/or peritoneal effusion (e.g., effusion affecting normal organ function and/or requiring percutaneous drainage or diuretic control);
  * autoimmune disease requiring chronic steroid use;
  * prior history of a stroke or transient ischemic attack within the last 6 months;
  * history of significant cardiac disease within 6 months prior to starting treatment such as myocardial infarction, unstable angina, cardiomyopathy, congestive heart failure;
  * prior allogeneic stem cell transplantation or organ transplantation.
* Central nervous system metastases

  * Symptomatic uncontrolled brain metastases requiring corticosteroid treatment.
  * History of spinal cord compression unless after definitive treatment the patient has clinically stable disease (SD) for at least 28 days prior to starting investigational agent(s).
* Pregnant or lactating (breastfeeding) women.
* Patients receiving concurrent treatment with other anti-cancer therapy or other investigational anti-cancer agents.
* Active or prior documented autoimmune or inflammatory disorders, including: inflammatory bowel disease (e.g. colitis or Crohn's disease), diverticulitis with the exception of diverticulosis, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea, systemic lupus erythematosus, Sarcoidosis syndrome, Wegener syndrome (granulomatosis with polyangiitis), rheumatoid arthritis, hypophysitis, uveitis, etc., within the past 3 years prior to the start of treatment.
* Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune conditions only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions considered to be of low risk for recurrence are permitted to enroll.
* Patients must not have been administered a live vaccine ≤ 4 weeks before enrollment.

Note: Seasonal vaccines for influenza are general inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and not allowed.

* QTc (using the Fridericia correction calculation) >470 msec or >450 msec if history of additional risk factors for Torsade de Pointe (e.g. heart failure, hypokalemia, family history of Long QT Syndrome) or use of concomitant medications that prolong the QT/QTc interval.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To efficiently identify based on objective response rate (ORR), by investigator assessment using RECIST 1.1, promising immunotherapy combinations for the treatment of high grade serous ovarian cancer for later validation in randomized trials | 36 months

SECONDARY OUTCOMES:
Evaluate ORR by investigator assessment using RECIST 1.1 | 36 months
Determine progression-free survival of immunotherapy regimens (RECIST 1.1 and iRECIST) | 36 months
Determine overall-survival of immunotherapy regimens (RECIST 1.1 and iRECIST) | 36 months
Number and severity of adverse events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Helen MacKay, Study Chair — Sunnybrook Health Sciences Centre, Toronto, Ontario Canada; Anna Tinker, Study Chair — BCCA - Vancouver Cancer Centre, BC Canada
Locations (7):
- The University of Chicago Medical Center, Chicago, Illinois, United States
- Canada (6):
  - BCCA - Kelowna, Kelowna, British Columbia
  - BCCA - Vancouver, Vancouver, British Columbia
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No